CLINICAL TRIAL: NCT05765084
Title: Integration of the PD-L1 Inhibitor Atezolizumab and WT1/DC Vaccination Into Platinum/Pemetrexed-based First-line Treatment for Epithelioid Malignant Pleural Mesothelioma
Acronym: Immuno-MESODEC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Algemeen Ziekenhuis Maria Middelares (Other); Vitaz (Other); Kom Op Tegen Kanker (Other); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCRG21-001
Record Dates: First submitted 2023-02-13; First posted 2023-03-13 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: Dendritic cell vaccination; Chemo-immunotherapy; Wilms' Tumor 1 (WT1); Checkpoint inhibition
MeSH Terms: conditions — Mesothelioma, Malignant; Wilms Tumor | interventions — atezolizumab; Platinum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm (Experimental): Standard of care chemotherapy, complemented with atezolizumab and WT1/DC vaccination
  Interventions: Biological: Dendritic cell vaccination; Drug: Atezolizumab; Drug: Platinum/pemetrexed based chemotherapy

INTERVENTIONS:
Biological: Dendritic cell vaccination — WT1/DC vaccines (8-10 x 10^6 cells in 500 μL saline solution with 5% human albumin) will be administered through intradermal injection at 5 sites (100 μL/site) in the ventromedial region of the upper arm (5-10 cm from the axillary lymph nodes). Injection sites will alternate between left and right arms. WT1/DC vaccines are administered on day 14 of each 3-weekly platinum/pemetrexed-based chemotherapy cycle. Additional WT1/DC vaccinations after the study treatment schedule can be administered (optional) at 4-weekly intervals (± 1 week).
Drug: Atezolizumab — Atezolizumab (1200 mg) will be administered on day 0 of each 3-weekly platinum/pemetrexed-based chemotherapy cycle. Atezolizumab should be administered before chemotherapy administration as an IV infusion over 60 (±15) minutes. If the first infusion is tolerated, all subsequent infusions may bedelivered over 30 (±10) minutes. Additional atezolizumab treatment (1680 mg) after the study treatment schedule can be administered (optional) at 4-weekly intervals (± 1 week) as an IV infusion over 30-60 minutes.
Drug: Platinum/pemetrexed based chemotherapy — On the first day of each cycle (day 0), pemetrexed 500 mg/m2 should be administered as intravenous (IV) infusion over 10 minutes, followed by cisplatin 75 mg/m2 as IV over approximately 2 hours. The actual doses of the drugs to be administered to patients will be determined by calculating the patient's body surface area at the beginning of each cycle. For ease of dose administration, the protocol allows ± 5% variance in the calculated total dose per infusion. If deemed necessary, the treating physician can decide to replace cisplatin by carboplatin. In that case, carboplatin will be delivered to an area under the concentration-time curve (AUC) of 5 as an IV infusion over 1 hour.

SUMMARY:
In this multicenter phase I/II trial, the programmed death-ligand 1 (PD-L1) inhibitor atezolizumab and dendritic cells (DCs) loaded with the mesothelioma-associated tumor antigen WT1 will be integrated into platinum/pemetrexed-based first-line chemotherapy for the treatment of epitheloid malignant pleural mesothelioma (MPM). The general objective is to provide the first-in-human experimental demonstration that the combination of platinum/pemetrexed-based chemotherapy with atezolizumab and WT1/DC vaccination is feasible and safe, has clinical activity and enables the induction of mesothelioma-specific immune responses in patients with MPM.

DETAILED DESCRIPTION:
Malignant pleural mesothelioma (MPM) is a highly aggressive and in virtually all cases fatal cancer that is tightly associated with prior asbestos exposure. Despite some improvement over time, the prognosis of patients diagnosed with MPM remains dismal with a median overall survival from diagnosis of only 9-16 months.

In this single arm phase I/II trial the investigators want to demonstrate the feasibility and safety of integrating the programmed death-ligand 1 (PD-L1) inhibitor atezolizumab and WT1-targeted dendritic cell vaccination in epitheloid MPM patients in conjunction with first line platinum/pemetrexed-based chemotherapy. In addition, chemo-immunotherapy-induced immunogenicity will be studied and patient's clinical outcome will be documented for comparison with current patient's outcome allowing indication of the added value.

Fifteen patients diagnosed with histologically proven epithelial MPM (stage I-IV) will be included. Patients should be able to undergo leukapheresis, chemotherapy and immunotherapy. Patients who underwent prior treatment for MPM or with a history of another malignancy within the last three years will be excluded.

The intention of this study is to administer four 3-weekly (±3 days) platinum/pemetrexed-based chemotherapy cycles (CT1-4) combined with atezolizumab treatments (A1-4) and autologous WT1 messenger (m)RNA-loaded dendritic cells (V1-4) at day 0 and day 14 (±3 days) of each chemotherapy cycle, respectively.

Additional atezolizumab doses and/or WT1/DC vaccines after the chemo-immunotherapy study scheme can be administered to the patient if consent for continuation of atezolizumab treatment and/or WT1/DC vaccination was obtained and residual WT1/DC vaccine aliquots are available. In that case, atezolizumab and/or WT1/DC vaccines will be administered on a 4-weekly basis (±1 week). The WT1/DC vaccines will be administered within 1 week after atezolizumab administration.

After the final WT1/DC vaccination and/or atezolizumab administration, patients will enter a follow-up phase that lasts for up to 90 days after final WT1/DC vaccination and/or atezolizumab administration or 24 months after diagnosis, whichever occurs later.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the following criteria to be eligible to participate in the study:

* Signed informed consent
* Diagnosis with histologically proven epithelioid unresectable MPM (stage I-IV)
* Age ≥ 18 years at the time of signing informed consent
* World Health Organization (WHO) performance status 0-1
* Adequate hematologic and end-organ function, defined by the following laboratory test results, obtained at the time of screening:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L (1500/μL) without granulocyte colony- stimulating factor support
  * Lymphocyte count ≥ 0.5 x 10^9/L (500/μL)
  * Platelet count ≥ 100 x 10^9/L (100,000/μL) without transfusion
  * Hemoglobin ≥ 90 g/L (9 g/dL) Patients may be transfused to meet this criterion
  * Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤ 2.5 x upper limit of normal (ULN), with the following exceptions:
  * Patients with documented liver metastases: AST and ALT ≤ 5 x ULN
  * Patients with documented liver or bone metastases: ALP ≤ 5 x ULN
  * Total bilirubin ≤ 1.5 x ULN with the following exception:
  * Patients with known Gilbert disease: total bilirubin ≤ 3 x ULN
  * Creatinine ≤ 1.5 x ULN
  * Albumin ≥ 25 g/L (2.5 g/dL)
  * For patients not receiving therapeutic anticoagulation: prothrombin international normalized ration (PT-INR) and activated partial thromboplastin time (APTT) ≤ 1.5 x ULN
* Negative Human Immunodeficiency Virus (HIV) test at screening
* Negative hepatitis B surface antigen (HBsAg) test at screening
* Negative total hepatitis B core antibody (HBcAb) test at screening, or positive total HBcAb test followed by a negative hepatitis B virus (HBV) DNA test at screening

  * The HBV DNA test will be performed only for patients who have a negative HBsAg test and a positive total HBcAb test.
* Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening. The HCV RNA test must be performed for patients who have a positive HCV antibody test.
* Willing and able to comply with the study protocol, as judged by the treating physician
* Women of childbearing potential must have a negative serum or urine pregnancy test at the time of screening and agree to use effective contraception (<1% failure rate per year) before, during and for at least five months after the last atezolizumab administration or at least hundred days after the last WT1/DC vaccine administration (whichever takes longer). Men must agree to use effective contraception before, during and for at least hundred days after the last study treatment administration.

Exclusion Criteria:

Subjects who fulfill any of the following criteria will not be eligible for admission into the study:

* History of malignancy within 3 years prior to initiation of study treatment, with the exception of the cancer under investigation in this study and malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate > 90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer
* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases. Asymptomatic patients with treated CNS lesions are eligible, provided that all of the following criteria are met:

  * Measurable disease, per RECIST v1.1, must be present outside the CNS.
  * The patient has no history of intracranial hemorrhage or spinal cord hemorrhage.
  * The patient has not undergone stereotactic radiotherapy within 7 days prior to initiation of study treatment, whole-brain radiotherapy within 14 days prior to initiation of study treatment, or neurosurgical resection within 28 days prior to initiation of study treatment.
  * The patient has no ongoing requirement for corticosteroids as therapy for CNS disease.
  * If the patient is receiving anti-convulsant therapy, the dose is considered stable.
  * Metastases are limited to the cerebellum or the supratentorial region (i.e., no metastases to the midbrain, pons, medulla, or spinal cord).
  * There is no evidence of interim progression between completion of CNS directed therapy and initiation of study treatment.
  * Asymptomatic patients with CNS metastases newly detected at screening are eligible for the study after receiving radiotherapy and/or surgery, with no need to repeat the screening brain scan.
* History of leptomeningeal disease
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, anti-phospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions:

  * Patients with a history of autoimmune-related hypothyroidism who are on thyroid replacement hormone are eligible for the study.
  * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
  * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

    * Rash must cover < 10% of body surface area
    * Disease is well controlled at baseline and requires only low-potency topical corticosteroids
    * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids within the previous 12 months.
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina
* Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
* Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia, or any active infection that could impact patient safety
* Prior treatment for MPM
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment. Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease (COPD) exacerbation) are eligible for the study.
* Prior allogeneic stem cell or solid organ transplantation
* Use of any investigational agent within 28 days before study enrollment
* Pregnant or breastfeeding. Female subjects who are breastfeeding should discontinue nursing prior to the first dose of study treatment and until at least hundred days after the last study treatment administration.
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the final dose of atezolizumab.
* Current treatment with anti-viral therapy for HBV
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
* Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor-α [TNF-α] agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

  * Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) may be eligible for the study after Medical Monitor confirmation has been obtained.
  * Patients who received mineralocorticoids (e.g., fludrocortisone), inhaled or low dose corticosteroids for COPD or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
* Treatment with systemic immunostimulatory agents (including but not limited to interferons or interleukin-2) within 4 weeks or 5 drug-elimination half-lives of the drug, whichever is longer, prior to initiation of study treatment
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation
* Any other condition, either physical or psychological, or reasonable suspicion thereof on clinical or special investigation, which contraindicates the use of atezolizumab, pemetrexed, cisplatin/carboplatin and/or WT1/DC vaccination, or may negatively affect patient compliance, or may place the patient at higher risk of potential treatment complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-02-24 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients that experienced (S)AEs possibly, probably or definitely related to pemetrexed and/or cisplatin/carboplatin and/or atezolizumab and/or WT1/DC vaccination | through study completion, an average of 2 years
  The relationship of an AE to the investigational agents will be determined by the Investigator as either related or non-related, based on their clinical judgment.
Number and grade of AEs and SAEs | through study completion, an average of 2 years
  AEs are defined and graded according to the latest version of the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) and Common Toxicity Criteria (CTC)
Proportion of patients who completed study treatment schedule | After the chemoimmunotherapy treatment (+/- 18 weeks after entry to trial)
  Study treatment schedule = administration of four platinum/pemetrexed-based chemotherapy cycles (CT1-4) in combination with four atezolizumab treatments (A1-4) and four WT1/DC vaccinations (V1-4).

SECONDARY OUTCOMES:
Best overall response | through study completion, an average of 2 years
  Best overall response will be determined per patient as the best overall response designation. The BOR categories are complete response (CR), partial response (PR), stable disease (SD) and progressive disease (PD).
Duration of response | through study completion, an average of 2 years
  Duration of response will be calculated for patients with an objective response as the time between the first date of the first documented tumor response (CR or PR) and the subsequent date of the objectively documented disease progression or death, whichever occurs first, or the last tumor assessment in case of censoring.
Disease control rate | through study completion, an average of 2 years
  Disease control rate is defined as the proportion of patients whose BOR is either CR, PR or SD, where the dominator is the total number of evaluable patients.
Objective response rate | through study completion, an average of 2 years
  Objective response rate is defined as the proportion of patients whose BOR is either CR or PR, where the dominator is the total number of evaluable patients.
Progression-free survival | through study completion, an average of 2 years
  Progression-free survival is defined as the time (in months) between start of the platinum/pemetrexed-based chemotherapy treatment and the date of progression or death due to any cause, whichever occurs first. At the time of analysis, patients without a recorded event will be censored at the time of the last objective disease assessment.
Overall survival | through study completion, an average of 2 years
  Overall survival is defined as the time (in months) between diagnosis/start of treatment and death due to any cause. At the time of analysis, patients without a recorded event will be censored at the time they were last known to be alive.
Functional WT1-specific T cell responses | After the fourth DC vaccine, at the time of disease progression (if applicable) and 12 months after the start of 1L chemo-immunotherapy in case of sustained disease control
  Change in the proportion of T cells exhibiting functional WT1-specific T cell responses as measured by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Zwi N Berneman, MD, PhD, Study Director — Antwerp University Hospital, Division of Hematology and Center for Cell Therapy and Regenerative Medicine; Paul Germonpré, MD, PhD, Principal Investigator — AZ Maria Middelares, Respiratory Oncology & Integrated Cancer Center Ghent; Koen Deschepper, MD, Principal Investigator — VITAZ, Division of Pulmonary and Infectious Diseases
Locations (3):
- Belgium (3):
  - Antwerp University Hospital, Edegem, Antwerp
  - AZ Maria Middelares, Ghent
  - VITAZ, Sint-Niklaas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Van Tendeloo VF, Van de Velde A, Van Driessche A, Cools N, Anguille S, Ladell K, Gostick E, Vermeulen K, Pieters K, Nijs G, Stein B, Smits EL, Schroyens WA, Gadisseur AP, Vrelust I, Jorens PG, Goossens H, de Vries IJ, Price DA, Oji Y, Oka Y, Sugiyama H, Berneman ZN. Induction of complete and molecular remissions in acute myeloid leukemia by Wilms' tumor 1 antigen-targeted dendritic cell vaccination. Proc Natl Acad Sci U S A. 2010 Aug 3;107(31):13824-9. doi: 10.1073/pnas.1008051107. Epub 2010 Jul 14. PMID 20631300
- [Background] Anguille S, Van de Velde AL, Smits EL, Van Tendeloo VF, Juliusson G, Cools N, Nijs G, Stein B, Lion E, Van Driessche A, Vandenbosch I, Verlinden A, Gadisseur AP, Schroyens WA, Muylle L, Vermeulen K, Maes MB, Deiteren K, Malfait R, Gostick E, Lammens M, Couttenye MM, Jorens P, Goossens H, Price DA, Ladell K, Oka Y, Fujiki F, Oji Y, Sugiyama H, Berneman ZN. Dendritic cell vaccination as postremission treatment to prevent or delay relapse in acute myeloid leukemia. Blood. 2017 Oct 12;130(15):1713-1721. doi: 10.1182/blood-2017-04-780155. Epub 2017 Aug 22. PMID 28830889
- [Background] Van Tendeloo VF, Ponsaerts P, Lardon F, Nijs G, Lenjou M, Van Broeckhoven C, Van Bockstaele DR, Berneman ZN. Highly efficient gene delivery by mRNA electroporation in human hematopoietic cells: superiority to lipofection and passive pulsing of mRNA and to electroporation of plasmid cDNA for tumor antigen loading of dendritic cells. Blood. 2001 Jul 1;98(1):49-56. doi: 10.1182/blood.v98.1.49. PMID 11418462
- [Background] Smits EL, Anguille S, Cools N, Berneman ZN, Van Tendeloo VF. Dendritic cell-based cancer gene therapy. Hum Gene Ther. 2009 Oct;20(10):1106-18. doi: 10.1089/hum.2009.145. PMID 19656053
- [Background] Benteyn D, Anguille S, Van Lint S, Heirman C, Van Nuffel AM, Corthals J, Ochsenreither S, Waelput W, Van Beneden K, Breckpot K, Van Tendeloo V, Thielemans K, Bonehill A. Design of an Optimized Wilms' Tumor 1 (WT1) mRNA Construct for Enhanced WT1 Expression and Improved Immunogenicity In Vitro and In Vivo. Mol Ther Nucleic Acids. 2013 Nov 19;2(11):e134. doi: 10.1038/mtna.2013.54. PMID 24253259
- [Background] Versteven M, Van den Bergh JMJ, Marcq E, Smits ELJ, Van Tendeloo VFI, Hobo W, Lion E. Dendritic Cells and Programmed Death-1 Blockade: A Joint Venture to Combat Cancer. Front Immunol. 2018 Mar 1;9:394. doi: 10.3389/fimmu.2018.00394. eCollection 2018. PMID 29599770
- [Background] Van den Bergh JMJ, Smits ELJM, Berneman ZN, Hutten TJA, De Reu H, Van Tendeloo VFI, Dolstra H, Lion E, Hobo W. Monocyte-Derived Dendritic Cells with Silenced PD-1 Ligands and Transpresenting Interleukin-15 Stimulate Strong Tumor-Reactive T-cell Expansion. Cancer Immunol Res. 2017 Aug;5(8):710-715. doi: 10.1158/2326-6066.CIR-16-0336. Epub 2017 Jun 21. PMID 28637876
- [Background] Versteven M, Van den Bergh JMJ, Broos K, Fujiki F, Campillo-Davo D, De Reu H, Morimoto S, Lecocq Q, Keyaerts M, Berneman Z, Sugiyama H, Van Tendeloo VFI, Breckpot K, Lion E. A versatile T cell-based assay to assess therapeutic antigen-specific PD-1-targeted approaches. Oncotarget. 2018 Jun 12;9(45):27797-27808. doi: 10.18632/oncotarget.25591. eCollection 2018 Jun 12. PMID 29963238
- [Background] Van Driessche A, Berneman ZN, Van Tendeloo VF. Active specific immunotherapy targeting the Wilms' tumor protein 1 (WT1) for patients with hematological malignancies and solid tumors: lessons from early clinical trials. Oncologist. 2012;17(2):250-9. doi: 10.1634/theoncologist.2011-0240. Epub 2012 Jan 30. PMID 22291091
- [Background] Anguille S, Smits EL, Lion E, van Tendeloo VF, Berneman ZN. Clinical use of dendritic cells for cancer therapy. Lancet Oncol. 2014 Jun;15(7):e257-67. doi: 10.1016/S1470-2045(13)70585-0. PMID 24872109
- [Derived] Van den Bossche J, De Laere M, Deschepper K, Germonpre P, Valcke Y, Lamont J, Stein B, Van Camp K, Germonpre C, Nijs G, Roelant E, Anguille S, Lion E, Berneman Z. Integration of the PD-L1 inhibitor atezolizumab and WT1/DC vaccination into standard-of-care first-line treatment for patients with epithelioid malignant pleural mesothelioma-Protocol of the Immuno-MESODEC study. PLoS One. 2024 Jul 15;19(7):e0307204. doi: 10.1371/journal.pone.0307204. eCollection 2024. PMID 39008481